CLINICAL TRIAL: NCT04721626
Title: A Topical Antiseptic Bundle for Decreasing Surgical Site Infection in Head and Neck Cancer Patients: Perioperative Effects on the Oral Microbiome
Brief Title: Topical Antisepsis in Head and Neck Cancer Surgery
Status: Completed | Type: Observational
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Joseph Zenga, Assistant Professor, Medical College of Wisconsin
Other Study IDs: PRO00039230
Record Dates: First submitted 2021-01-19; First posted 2021-01-22 (Actual); Last update posted 2022-02-07 (Actual); Status verified 2022-02

CONDITIONS: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — chlorhexidine gluconate; Povidone-Iodine; Minocycline

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Swabs will be taken of the mouth, nose, surgical site and environment. Recombinant 16s DNA (16 s) sequencing will be used to identify bacteria present at those sites.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Chlorhexidine Gluconate — Preoperative: The patient's dentition, or mandibular alveolus in the absence of dentition, will be brushed for two minutes with 0.12% chlorhexidine gluconate.
  Intraoperative: The wound will be irrigated for 60 seconds with 0.05% chlorhexidine after it is irrigated with povidone-iodine.
  Postoperative: Patients will swish and spit/suction 15mL 0.12% Chlorhexidine Gluconate (CHG) oral rinses for 30 seconds every six hours for two days (8 total administrations)
  Other Names: Peridex
Drug: Povidone-iodine — Preoperative: The oral cavity and oropharyngeal mucosa as well as the nasal vestibules will be coated with 5% povidone-iodine which will stand for at least three minutes prior to incision.
  Intraoperative: The wound will be irrigated for 60 seconds with 10% povidone-iodine.
  Other Names: Iodopovidone
Drug: Tetracycline Ointment — Postoperative: ~10g 3% tetracycline ointment will be placed into the oral cavity to coat the dorsal tongue and any oral suture lines every six hours for two days (8 total doses).
  Other Names: Adoxa CK; Adoxa TT; Amzeeq; Cleeravue-M; Zilxi

SUMMARY:
This is a single-arm prospective trial of an intra- and postoperative topical antiseptic bundle. The study will recruit patients undergoing an open surgical resection of the upper aerodigestive tract requiring a planed vascularized reconstruction, which may be either pedicled and/or free flap. The objectives are to evaluate antimicrobial effects of a perioperative topical antiseptic bundle and to identify the source of surgical site infection as well as the rate of 30-day adverse events in head and neck cancer.

DETAILED DESCRIPTION:
The study design is a single-arm prospective trial. It will investigate the microbial effects of topical antisepsis on upper aerodigestive tract and reconstructive surgery in head and neck cancer patients. The primary hypothesis is that topical antisepsis will significantly decrease oral bacterial load and the presence of pathogenic organisms. Secondary outcomes will include identification of the source of the infectious bacterial organisms, surgical and non-surgical site infections, serious topical antisepsis-related complications, serious adverse events, and hospital revisits. The study populations will include head and neck cancer patients age 18 or greater undergoing head and neck reconstructive surgery in which there is a communication between the upper aerodigestive tract and the cervical skin which requires a planned vascularized reconstruction, either a regional pedicled flap or a free tissue transfer. The accrual goal will be 25 patients. Data collection will occur in both the inpatient and outpatient settings. Patients will be enrolled during their preoperative clinic visit. Each patient will be followed for study outcomes until 30 days postoperatively.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older.
2. Planned to undergo an open surgical procedure requiring a communication between the upper aerodigestive tract and cervical skin with a planned vascularized reconstruction, which may be either a regional pedicled and/or free flap.
3. Subsites reconstructed must include at least one of the following: oral cavity, oropharynx, larynx, hypopharynx, and/or cervical esophagus.
4. Eligible patients must be undergoing surgery related to treatment for head and neck cancer. This includes immediate reconstruction after tumor ablation as well as reconstruction for delayed cancer-related indications including radionecrosis or improvement in functional outcomes after head and neck cancer treatment.
5. Voluntary written consent must be given before performance of any study-related procedure not part of standard medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to future medical care.

Exclusion Criteria:

1. True allergy to any study-related medications
2. Active infection at the time of surgery
3. Pregnancy or actively breastfeeding mothers. Female subjects who are both lactating and breastfeeding or of childbearing potential who have a positive serum test during screening.
4. Patients incarcerated in state or federal penitentiaries
5. Patients with a serious medical or psychiatric illness likely to interfere with participation in this clinical study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligibility: Patients ≥ 18 years old planned to undergo surgical resection of the upper aerodigestive tract for a cancer-related indication and requiring reconstruction which may be either a regional pedicled and/or free tissue transfer.
Sampling Method: Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2021-01-06 (Actual); Primary Completion 2021-05-28 (Actual); Study Completion 2021-10-04 (Actual)

PRIMARY OUTCOMES:
Oral microbial abundance in preoperative samples measured by quantitative bacteriology. | Baseline (immediately preoperative)
  Bacteria will be measured as colony forming unit/mL.
Oral microbial abundance in preoperative samples measured by 16s sequencing. | Baseline (immediately preoperative)
  This will be measured by the number of operational taxonomic units.
Oral microbial abundance in intraoperative samples prior to antiseptic irrigations measured by quantitative bacteriology. | During surgery before wound irrigation
  Bacteria will be measured as colony forming unit/mL.
Oral microbial abundance in intraoperative samples prior to antiseptic irrigations measured by 16s sequencing. | During surgery before wound irrigation
  This will be measured by the number of operational taxonomic units.
Oral microbial abundance in samples after intraoperative antiseptic irrigations measured by quantitative bacteriology. | During surgery following wound irrigation
  Bacteria will be measured as colony forming unit/mL.
Oral microbial abundance in samples after intraoperative antiseptic irrigations measured by 16s sequencing. | During surgery following wound irrigation
  This will be measured by the number of operational taxonomic units.
Oral microbial abundance in postoperative samples measured by quantitative bacteriology. | Postoperative day 3.
  Bacteria will be measured as colony forming unit/mL.
Oral microbial abundance in postoperative samples measured by 16s sequencing. | Postoperative day 3.
  This will be measured by the number of operational taxonomic units.

SECONDARY OUTCOMES:
The number of subjects with surgical site infection | 30 days
  Surgical site infection diagnosis must be performed by the attending physician and occur within 30 days post-operatively. Diagnosis will include either: 1) purulent drainage from incision, 2) incision spontaneously dehisced or opened by the surgeon because of infection, 3) abscess or other evidence of infection involving a deep incision; or 4) surgical site infection diagnosis by the surgeon.
Number of subjects with 30-day hospital revisits | Up to 30 days
  Defined as any unanticipated hospital readmission within 30 days of the index surgery.
Number of subjects with non-surgical site infections | 30 days
  An infection of the tracheobronchial tree, urinary tract, or blood, as determined by the isolation of pathogenic microorganisms from these sites in the setting of clinical signs and symptoms of infection in accordance with the International Nosocomial Infection Control Consortium (INICC) criteria. Pneumonia, clinical sepsis, and symptomatic urinary tract infection without an identified pathogenic microorganism may be diagnosed according to the INICC guidelines.
The number of subjects with serious topical antisepsis-related complications | 30 days
  Serious adverse event is deemed related to or probably related to the topical antiseptic agent. When topical antiseptic-related complications are suspected by the attending physician, the infectious disease service will be consulted, and a serious topical antiseptic-related complication will be diagnosed based on their recommendations.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Zenga, MD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Froedtert Hospital & the Medical College of Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No